CLINICAL TRIAL: NCT00754234
Title: Iron Bioavailability From MyPyramid Menus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GFHNRC003
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Nonheme Iron Absorption
Keywords: iron absorption; iron requirements; dietary guidelines; MyPyramid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MyPyramid Menu Days 1-7 (Experimental): Iron absorption measured from one of the 7 different USDA MyPyramid menus for 1 day each, in randomized order for each subject, separated by 2 weeks
  Interventions: Behavioral: My Pyramid menu days 1, 2, 3, 4, 5, 6 or 7

INTERVENTIONS:
Behavioral: My Pyramid menu days 1, 2, 3, 4, 5, 6 or 7 — Iron absorption measured from one of seven different menus fed for 1 day each, in randomized order for each subject, with feedings separated by 2 weeks

SUMMARY:
This study will measure nonheme iron absorption from each of the 7 daily MyPyramid menus. Such measurements will confirm whether modifications are needed to meet dietary iron recommendations and will provide data useful for validation algorithms to calculate dietary iron bioavailability.

DETAILED DESCRIPTION:
Nonheme iron absorption is measured with 59Fe tracer added to a 1-day menu, with iron retention detected two weeks later in a whole body scintillation counter. Each subject has iron absorption measured from each of 7 1-d menus formulated to meet the US dietary guidelines (MyPyramid menus), with the order of menus randomly assigned. Each subject participates for 14 wk to test all 7 menus.

ELIGIBILITY:
Inclusion Criteria:

* Women 21 to 50 years old

Exclusion Criteria:

* Anemia,
* High blood pressure,
* Disorders affecting iron absorption or retention,
* Underlying medical conditions,
* Taking medication other than birth control pills or hormone replacement therapy,
* Pregnancy,
* Daily use of analgesics

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet R Hunt, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from the Grand Forks, North Dakota community in September 2007.
Pre-assignment Details: 154 applied,(47 applied too late, 30 did not meet inclusion criteria and 52 refused participation) 25 screened,4 excluded (3 did not pass screen and 1 refused participation), 5 alternates
Groups:
- MyPyramid Menus: USDA MyPyramid menus for Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
Period: Overall Study
Arm/Group | MyPyramid Menus
Started | 16 (7 Menus were consumed in randomized order)
Completed | 13 (2 participants did not receive the Day 1,4,5,6 menu and 1 did not receive the Day 2 menu)
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | MyPyramid Menus
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Nonheme Iron Absorption
Description: Absorption was estimated from whole body retention of a Iron-59 radiotracer, 2 weeks after consuming a menu labeled with the isotope, then normalized to a ferritin of 15 nanogram/milliLiter (ng/mL)
Time Frame: 2 weeks (wks)
Population: Analysis was per protocol
Measure: Log Mean (Standard Deviation); unit: percentage of nonheme Iron absorbed
Groups:
- MyPyramid Menu: USDA MyPyramid menus for Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
Arm/Group | MyPyramid Menu
Number analyzed (Participants) | 14
percentage of nonheme Iron absorbed | 2.31 (0.61)

ADVERSE EVENTS:
Arm/Group | MyPyramid Menus
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No